CLINICAL TRIAL: NCT01057732
Title: The Effect of Parathyroidectomy on Cardiovascular Risk Factors in Patients With Primary Hyperparathyroidism
Brief Title: Effects of Parathyroidectomy on Cardiovascular Risk Factors in Primary Hyperparathyroidism
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Avraham Ishay, Haemek Medical Center, Afula, Israel
Other Study IDs: 3630405
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2010-01

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- primary hyperparathyroidism: patients with primary hyperparathyroidism
- controls: subjects without primary hyperparathyroidism

SUMMARY:
Primary hyperparathyroidism (PHPT) is associated with increased cardiovascular morbidity. The benefit of surgical treatment in this respect is unclear.

This study was performed to evaluate the impact of parathyroidectomy (PTX) on cardiovascular risk profile.

DETAILED DESCRIPTION:
Patients with primary hyperparathyroidism (PHPT) have been shown to have an increased morbidity and mortality mainly due to cardiovascular disease. The precise mechanism of cardiovascular disease in PHPT is not well understood and probably multifactorial. Functional or structural alterations of vascular endothelial and smooth muscle cells may impair the vascular reactivity and lead to accelerated atherogenesis. Several cardiovascular risk factors such as obesity, hypertension, insulin resistance and hyperlipidemia are more prevalent in PHPT compared with controls.Patients with severe form of PHPT had a greater probability of metabolic syndrome (MS) and insulin resistance than patients with mild PHPT and eucalcemic subjects. Although the excess in cardiovascular mortality is significantly and independently related to serum calcium, the connection between the biochemical disturbances and the cardiovascular disorders in PHPT patients is not necessarily a cause-and-effect relationship. Indeed, the impact of surgical cure of hyperparathyroidism on cardiovascular risk factors and mortality is controversial. Some studies suggest that hypertension, dyslipidemia, and derangement of glucose metabolism improve after removal of overactive parathyroid tissue. Others have shown that cardiovascular risk markers remained unaltered after parathyroidectomy (PTX).

The aim of this study was to evaluate whether successful PTX is associated with decreased cardiovascular risk. We investigated indices of metabolic syndrome and insulin resistance as well as various cardiovascular risk factors in patients with manifest PHPT before and one year after successful PTX.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary hyperparthyroidism

Exclusion Criteria:

* Individuals with known diabetes mellitus,coronary heart disease, stroke

Ages: 18 Years to 80 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Primary hyperparathyroidism referred to Endocrine clinic. Controls recruited in community-based health centers.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2005-01; Primary Completion 2006-06 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrine Institute, Haemek Medical Center, Afula, Israel